CLINICAL TRIAL: NCT05210777
Title: Norms and Validation for IntelliSpace Cognition Spanish Version
Status: Completed | Type: Observational
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Collaborators: suAzio N.V. (Unknown)
Responsible Party: Sponsor
Other Study IDs: ICBE-S-000633
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Cognitive Functioning of Healthy Individuals; Hispanic
Keywords: Cognitive model; Cognitive assessment; Digital cognitive tests; Automated scoring; Algorithms
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: observation — no intervention

SUMMARY:
This study aims to validate and provide applicable norms for the United States (US) Spanish versions of the IntelliSpace Cognition (ISC) neuropsychological tests.

DETAILED DESCRIPTION:
The study will collect test scores from the Spanish speaking Hispanic US population for Spanish translations/adaptations of the ISC tests with the aim to assess how the Spanish language version of ISC tests compare to the English language version of ISC tests, and to create norms for the Spanish language version of the tests.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported:
* Participant is 18 years or older.
* Participant considers herself or himself to be Hispanic/Latino.
* Participant has Spanish as their primary and dominant language, or reports speaking Spanish as equally as good as she or he speaks English.
* Participant is able to see well (naturally or corrected by means of eyeglasses or lenses).
* Participant is able to hear well (naturally or corrected by means of a hearing aid).
* Participant is able to use their fingers, hands and arms to write symbols.
* Participant has valid health insurance.

Investigator observed:

* Participant is able to give informed consent.
* Participant is able to understand test instructions and participate fully in testing.
* Participant has normal fine and gross motor ability.

Exclusion Criteria:

* Self-reported:
* Participant has participated in previous studies where IntelliSpace Cognition was used (PJ-011726: "Study to establish the psychometric properties of the digital cognitive tests on the Philips IntelliSpace Cognition Platform" conducted during 2019 or ICBE-S-000233: "Norms Expansion and Validation for IntelliSpace Cognition" conducted during 2021).
* Participant is currently admitted to a hospital, assisted living, nursing home or a psychiatric facility.
* Participant is diagnosed with a neurological disorder or disease that may affect cognitive functioning (e.g., Parkinson's, brain tumor, stroke, Traumatic Brain Injury (TBI), epilepsy, encephalitis, dementia).

Admissible: Epilepsy with no more than 2 seizures and not currently receiving epilepsy treatment and not currently seeking medical attention related to seizures.

• Participant is diagnosed with a language disorder or aphasia (expressive or mixed receptive/expressive).

Admissible: Articulation disorder.

* Participant is diagnosed with a learning disorder.
* Participant is diagnosed with an autoimmune disorder that may affect cognitive functioning (e.g., LUPUS, Multiple Sclerosis).
* Participant is or was diagnosed with a current or past psychotic disorder (e.g., schizophrenia).
* Participant is diagnosed with a severe mood disorder. Admissible: Major Depressive Disorder in remission / Major Depressive Disorder with no current episode / Dysthymic Disorder / Adjustment Disorder
* Participant is diagnosed with a severe anxiety disorder. Admissible: Phobia / Anxiety disorders with symptoms not significant enough to interfere with test performance.
* Participant is or was diagnosed with current or past Autism Spectrum Disorder or Intellectual Disability.
* Participant is diagnosed with a current substance abuse or dependence. Admissible: In remission for at least 1 year.
* Participant has carried a substance abuse or dependence diagnosis for more than 10 years at any point in their life.
* Participant has an average alcohol consumption of 4 or more units per day.
* Participant uses medical marijuana.
* Participant uses recreational marijuana more than once a week.
* Participant uses recreational drugs other than alcohol and marijuana in the last 6 months (e.g., cocaine, ecstasy, LSD).
* Participant has been unconscious related to traumatic brain injury or "medical condition" for more than 20 minutes.

Admissible: Medication-induced or due to heat stroke.

* Participant has stayed in a hospital overnight due to a head injury.
* Participant has had a medical event requiring resuscitation in which they were non-responsive for more than 15 minutes.
* Participant has received chemotherapy treatment in the past 2 months.
* Participant has received electroconvulsive therapy (ECT).
* Participant has received radiation to the central nervous system.
* Participant experiences a physical condition or illness that interferes with normal cognitive functioning at work, school, Instrumental Activities of Daily Living (IADLs) etc.

Admissible: Diabetes, hypothyroidism, hypertension if controlled.

* Participant is currently taking anti-convulsants (e.g. Depakote, Lamictal or Lyrica, Gabapentin, Keppra, Topamax, Divalproex Sodium, Valproate Sodium, Levetiracetam, Lamotrigine, Pregabalin, Topiramate).
* Participant is currently taking anti-psychotics (e.g. Abilify, Rexulti, Zyprexa, Clozaril, Clozapine, Latuda, Seroquel, Risperdal, Risperidone, Aripipazle, Bexipiprazole, Olanzapine, Lurasidone HCL, Quetiapine).
* Participant is currently taking benzodiazepines (e.g. Diazepams, Valium, Klonopin, Ativan, Xanax, Lorazepam, Alprazolam, Clonazepam).
* Participant is currently taking psychostimulants (e.g. Amphetamines, Adderall, Ritalin, Methamphetamines, Dextroamphetamine, Methylphenidate HCL).

Admissible: Coffee.

* Participant is currently taking opioids (e.g. Oxycontin, Tramadol, Codeine, Dilaudid, Suboxone, Oxycodone, Percocet, Buprenorhine, Naloxone).
* Participant is currently taking antidepressants (e.g. Amitriptyline, Elavil, Pamelor, Tofranil, Vivactil, Imipramine, Protriptyline HCL).

Admissible: Antidepressants that are not tricyclic.

* Participant is currently taking oxybutynin (Ditropan).
* Participant is currently seeking medical diagnostic procedures for cognitive difficulties from a medical professional.
* Participant has received neuropsychological testing before. Admissible: Previous MMSE (-2) or MoCA testing more than 6 months prior.

Investigator observed:

* Participant shows evidence of current cognitive impairment.
* Participant displays disruptive behavior or insufficient compliance with testing to ensure a valid assessment.
* Participant is primarily nonverbal or uncommunicative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population is healthy Spanish-speaking adult participants from the US Hispanic subpopulation, with various sex, age, and education levels. All participants will be aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Validate the ISC Scores for Spanish Speaking population in US | Two months
  To collect test scores from Spanish speaking Hispanic US population for Spanish translations/adaptations of the ISC tests with the aim to assess how the Spanish language version of ISC tests compare to the English language version of ISC tests, and to create norms for the Spanish language version of the tests.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - suAzio, Hollywood, California
  - suAzio, Hollywood, Florida

IPD SHARING:
Plan to Share IPD: No